CLINICAL TRIAL: NCT01929694
Title: The Effect of Consuming a Guaraná and Vitamin and Mineral Complex Before a Morning Exercise Session on Affect, Exertion and Substrate Metabolism During Exercise and Cognitive Performance During the Post-exercise Recovery Period
Brief Title: The Effect of Consuming a guaraná and Vitamin/Mineral Complex Pre-exercise on Affect, Exertion, Metabolism and Cognition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 9B2
Record Dates: First submitted 2013-08-19; First posted 2013-08-28 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Affect and Exertion During and Post-exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Berocca Boost (Active Comparator): Guarana and vitamin and mineral complex, one tablet dissolved in 250ml water taken once.
  Interventions: Dietary Supplement: Berocca Boost
- Placebo (Placebo Comparator): Matched placebo tablet, one tablet dissolved in 250ml water taken once.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Berocca Boost
  Arms: Berocca Boost
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Consuming a guaraná and vitamin and mineral complex can improve mental fatigue and cognitive function at rest; guaraná also contains caffeine, which can reduce perceived exertion and increase fat burning during exercise. The purpose of this study is to test whether consuming a guaraná and vitamin and mineral product before exercise influences affect (mood), physical exertion and fat burning during exercise and mental fatigue, cognitive performance and affect post-exercise.

ELIGIBILITY:
Inclusion Criteria:

Individuals must be:

* Healthy
* Male
* Aged between 18 and 35years
* Habitually active (exercising at least twice a week)
* Able to run at a moderate pace for 30 minutes non-stop on a treadmill

Exclusion Criteria:

Individuals will not be eligible to take part in this study if they:

* have a history of neurological or psychiatric diseases excluding anxiety or depression
* have a current diagnosis of depression or anxiety
* have a history of significant head trauma, metabolic, endocrine or cardiac disorders
* have smoked within the last 3 months,
* have high blood pressure >140/90mmHg
* consume > 500 mg caffeine per day from all dietary sources
* have adverse reactions to caffeine containing products (i.e. tea, coffee, energy drinks, cola, Pepsi)
* are currently taking any pharmaceuticals
* have habitual taken dietary supplements within the last 4 weeks (defined as ≥3 consecutive days or ≥4 days in total per week)
* have current or history of drug or alcohol abuse
* have participated in another clinical trial within 30 days prior to screening
* have any condition which may interfere with your ability to perform assessments
* have any history of hypersensitivity to the investigational product or its active or inactive constituents or any food allergy or intolerance

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Affect | Assessed pre-exercise, at 10min intervals during exercise and 45 and 75min post-exercise
  Affect measured using the Feeling Scale and Felt Arousal Scale

SECONDARY OUTCOMES:
Exertion | Measured at 10min intervals during exercise
  Rate of perceived exertion measured using the Borg scale

OTHER OUTCOMES:
Cognitive Function | Assessed at baseline, pre-exercise and immeadiately and 75min post-exercise
  Participants will complete a set of cognitive tasks (Immediate Word Recall, Choice Reaction Time, Rapid visual information processing task, Numeric Working Memory, Delayed word Recall, Word Recognition and Picture Recognition) measuring episodic memory, working memory, attention and decision making.
Mood | Assessed at baseline, pre-exercise and immeadiately and 75min post-exercise
  Assessed using the Bond-Lader Visual Analogue Scales (VAS) and Energy VAS (concentration, physical stamina, mental stamina)
Substrate Metabolism | Measured at 10min intervals during exercise
  Measured using an online gas analysis system (Cortex). Oxygen uptake, carbon dioxide production, fat and carbohydrate oxidation and energy expenditure will be measured for 1 min at each 10min interval.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Veasey, MSc, Principal Investigator — Northumbria University
Locations (1):
- Brain, Performance and Nutrition Research Centre, Northumbria Univerity, Newcastle upon Tyne, Tyne and Wear, United Kingdom